CLINICAL TRIAL: NCT01423071
Title: Chronisch Obstruktive Lungenerkrankung Und Pulmonale Hypertonie: Prävalenz Und Lebensqualität
Brief Title: Chronic Obstructive Pulmonary Disease and Pulmonary Hypertension: Prevalence and Quality of Life
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Collaborators: Actelion Pharmaceuticals Deutschland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: WI_PH+COPD_73/2011
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Hypertension; Chronic obstructive pulmonary disease; Prevalence; Quality of life
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- COPD with PH: COPD patients with confirmed diagnosis of PH.
- COPD without PH: COPD patients without confirmed diagnosis of PH
- PAH without COPD: PAH patients who do not suffer from COPD

SUMMARY:
The purpose of this study is to determine the prevalence of pulmonary hypertension (PH) among patients suffering from Chronic Obstructive Pulmonary Disease (COPD) and to assess the quality of life in those patients with concomitant PH compared to COPD patients without PH and those only suffering from pulmonary arterial hypertension (PAH) respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Known or newly diagnosed COPD or PAH
* Written informed consent
* Present long-term oxygen treatment is no exclusion criterion

Exclusion Criteria:

* Age < 18 years
* Right-heart catheterization not reasonable
* Pregnancy, Lactation
* Life expectancy <12 months due to any diseases aside from COPD
* Any medical, psychological or other condition, which limits the patient's ability to provide informed consent
* No written informed consent provided
* Current participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In- and out-patients at the investigational center
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2011-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of PH | At baseline
  Prevalence of PH as defined by ESC/ERS guidelines (mean pulmonary arterial pressure ≥25 mmHg, assessed by right-heart catheterization) among the subgroup of COPD GOLD III and IV patients.

SECONDARY OUTCOMES:
Quality of life | One year
  Explorative data analysis to assess correlation between quality of life and PH, by comparison of COPD patients with and without PH and a reference group of patients with only PAH.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J Randerath, Prof. Dr. med., Principal Investigator — Wissenschaftliches Institut Bethanien e.V
Locations (1):
- Bethanien Hospital, Clinic for Pneumology and Allergology, Center for Sleep Medicine and Respiratory Care, Institute for Pneumology at the University Witten/Herdecke, Solingen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Warwick G, Thomas PS, Yates DH. Biomarkers in pulmonary hypertension. Eur Respir J. 2008 Aug;32(2):503-12. doi: 10.1183/09031936.00160307. PMID 18669790
- [Background] Kessler R, Faller M, Fourgaut G, Mennecier B, Weitzenblum E. Predictive factors of hospitalization for acute exacerbation in a series of 64 patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1999 Jan;159(1):158-64. doi: 10.1164/ajrccm.159.1.9803117. PMID 9872834
- [Background] Oswald-Mammosser M, Weitzenblum E, Quoix E, Moser G, Chaouat A, Charpentier C, Kessler R. Prognostic factors in COPD patients receiving long-term oxygen therapy. Importance of pulmonary artery pressure. Chest. 1995 May;107(5):1193-8. doi: 10.1378/chest.107.5.1193. PMID 7750305
- [Background] Barbera JA, Peinado VI, Santos S. Pulmonary hypertension in chronic obstructive pulmonary disease. Eur Respir J. 2003 May;21(5):892-905. doi: 10.1183/09031936.03.00115402. PMID 12765440
- [Background] Weitzenblum E. Chronic cor pulmonale. Heart. 2003 Feb;89(2):225-30. doi: 10.1136/heart.89.2.225. No abstract available. PMID 12527688
- [Background] Chaouat A, Bugnet AS, Kadaoui N, Schott R, Enache I, Ducolone A, Ehrhart M, Kessler R, Weitzenblum E. Severe pulmonary hypertension and chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 Jul 15;172(2):189-94. doi: 10.1164/rccm.200401-006OC. Epub 2005 Apr 14. PMID 15831842
- [Background] Arcasoy SM, Christie JD, Ferrari VA, Sutton MS, Zisman DA, Blumenthal NP, Pochettino A, Kotloff RM. Echocardiographic assessment of pulmonary hypertension in patients with advanced lung disease. Am J Respir Crit Care Med. 2003 Mar 1;167(5):735-40. doi: 10.1164/rccm.200210-1130OC. Epub 2002 Dec 12. PMID 12480614
- [Background] Burrows B, Kettel LJ, Niden AH, Rabinowitz M, Diener CF. Patterns of cardiovascular dysfunction in chronic obstructive lung disease. N Engl J Med. 1972 Apr 27;286(17):912-8. doi: 10.1056/NEJM197204272861703. No abstract available. PMID 5013974
- [Background] Weitzenblum E, Hirth C, Ducolone A, Mirhom R, Rasaholinjanahary J, Ehrhart M. Prognostic value of pulmonary artery pressure in chronic obstructive pulmonary disease. Thorax. 1981 Oct;36(10):752-8. doi: 10.1136/thx.36.10.752. PMID 7330793
- [Background] Vizza CD, Lynch JP, Ochoa LL, Richardson G, Trulock EP. Right and left ventricular dysfunction in patients with severe pulmonary disease. Chest. 1998 Mar;113(3):576-83. doi: 10.1378/chest.113.3.576. PMID 9515827
- [Background] Hoeper MM, Barbera JA, Channick RN, Hassoun PM, Lang IM, Manes A, Martinez FJ, Naeije R, Olschewski H, Pepke-Zaba J, Redfield MM, Robbins IM, Souza R, Torbicki A, McGoon M. Diagnosis, assessment, and treatment of non-pulmonary arterial hypertension pulmonary hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S85-S96. doi: 10.1016/j.jacc.2009.04.008. PMID 19555862
- [Background] Viegi G, Pistelli F, Sherrill DL, Maio S, Baldacci S, Carrozzi L. Definition, epidemiology and natural history of COPD. Eur Respir J. 2007 Nov;30(5):993-1013. doi: 10.1183/09031936.00082507. PMID 17978157
- [Background] Cenedese E, Speich R, Dorschner L, Ulrich S, Maggiorini M, Jenni R, Fischler M. Measurement of quality of life in pulmonary hypertension and its significance. Eur Respir J. 2006 Oct;28(4):808-15. doi: 10.1183/09031936.06.00130405. Epub 2006 May 17. PMID 16707511
- [Background] Hoeper MM, Oudiz RJ, Peacock A, Tapson VF, Haworth SG, Frost AE, Torbicki A. End points and clinical trial designs in pulmonary arterial hypertension: clinical and regulatory perspectives. J Am Coll Cardiol. 2004 Jun 16;43(12 Suppl S):48S-55S. doi: 10.1016/j.jacc.2004.02.010. PMID 15194178
- [Background] Rubenfire M, Lippo G, Bodini BD, Blasi F, Allegra L, Bossone E. Evaluating health-related quality of life, work ability, and disability in pulmonary arterial hypertension: an unmet need. Chest. 2009 Aug;136(2):597-603. doi: 10.1378/chest.08-1260. PMID 19666759
- [Background] McKenna SP, Doughty N, Meads DM, Doward LC, Pepke-Zaba J. The Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR): a measure of health-related quality of life and quality of life for patients with pulmonary hypertension. Qual Life Res. 2006 Feb;15(1):103-15. doi: 10.1007/s11136-005-3513-4. PMID 16411035
- [Background] McKenna SP, Ratcliffe J, Meads DM, Brazier JE. Development and validation of a preference based measure derived from the Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) for use in cost utility analyses. Health Qual Life Outcomes. 2008 Aug 21;6:65. doi: 10.1186/1477-7525-6-65. PMID 18718016
- [Background] Meads DM, McKenna SP, Doughty N, Das C, Gin-Sing W, Langley J, Pepke-Zaba J. The responsiveness and validity of the CAMPHOR Utility Index. Eur Respir J. 2008 Dec;32(6):1513-9. doi: 10.1183/09031936.00069708. Epub 2008 Sep 3. PMID 18768576